CLINICAL TRIAL: NCT00554255
Title: Phase I Study of SB751689 - Single and Multiple Oral Dose Study in Japanese Postmenopausal Women -
Brief Title: A Study of SB751689 in Japanese Postmenopausal Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 108543
Record Dates: First submitted 2007-11-02; First posted 2007-11-06 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Osteoporosis
Keywords: Pharmacodynamics; Japanese; safety; Pharmacokinetics
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: SB751689

SUMMARY:
To investigate the safety and tolerability, PK and PD of SB751689 following single and 5-day multiple oral doses of 100, 200, and 400 mg in Japanese postmenopausal subjects.

ELIGIBILITY:
Inclusion Criteria:

* The subject is considered as healthy by the investigator at screening.
* Healthy subjects are defined as individuals who are free from clinically significant illness or disease as determined by their medical history, physical examination, laboratory studies, and other tests
* Japanese healthy postmenopausal woman as defined as being amenorrheic for at least 1 year at screening with <157.79mIU/mL of FSH levels.
* Body weight >= 45 kg and BMI within the range 18.5 -25.0 kg/m2.
* The subject is within the following criteria as screening;Liver function tests (ALT, AST, GGT, alkaline phosphatase, total bilirubin), CPK, serum parathyroid hormone (iPTH) test, vitamin D (1,25(OH2 D3)) levels, Serum calcium
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Non-smokers (at least 6 months)
* The subject is able to attend all visits and complete the study.

Exclusion Criteria:

* The subject has any clinically relevant abnormality on medical examination, vital sign, clinical laboratory test or medical history at screening in the medical opinion of the investigator or the subject has a medical history that is not considered as eligible for inclusion in this study by the investigator.
* History of sensitivity to any of the study medications or components thereof (except pollenosis without any signs or symptoms).
* Participation in a clinical study or post-marketing study with an investigational or a non-investigational product or device within 4 months of preceding the first dose of study medication.
* Participation in another clinical study or post-marketing study in which the subject is or will be exposed to an investigational or a non-investigational product or device.
* Positive for syphilis, HIV antibody, hepatitis B antigen or hepatitis C antibody, HTLV-1 antibody at screening.
* Positive urine drug screen at screening.
* Donation of blood in excess of 400 mL within the previous 4 months or 200mL within the previous 1 month of screening.
* Use of prescription or non-prescription drugs, herbal and dietary supplements, within 14 days prior to the first dose of study medication.
* History of drug abuse or current conditions of drug abuse or alcoholism.
* History of regular alcohol consumption exceeding 7 units/week (>350mL of beer/unit) within 6 months of screening.
* Subjects with a history of renal, hepatic, or biliary disease.
* History of clinically significant cardiovascular disease.
* History of pernicious anemia, pancreatitis, osteosarcoma or kidney stones.
* Subjects who have had history of significant gastrointestinal disease (e.g., gastrointestinal malabsorptive disease, colostomy, chronic gastroesophageal reflux disease, Crohn's disease, ulcerative colitis, gastric or duodenal ulcer, gastrointestinal tract bleeding, short bowel syndrome, sprue, lactose intolerance, irritable bowel syndrome).
* Subjects with any history of a gastrointestinal surgical procedure that might affect the absorption of SB-751689 (e.g. cholecystectomy, gastrointestinal bypass surgery, partial or total gastrectomy, small bowel resection).
* Medical conditions which might alter bone metabolism, including hyperparathyroidism, hypoparathyroidism, hyperthyroidism, hypothyroidism, Paget's disease, malabsorption, or Cushing's syndrome, and hypogonadism, hypocalcemia, hypercalcemia, hypophosphatemia, hypomagnesemia, hypermagnesemia, osteopetrosis, osteomalacia, and recent (within one year) history of fracture or prolonged bedrest.

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2006-10-23; Study Completion 2006-12-12 (Actual)

PRIMARY OUTCOMES:
Adverse events, change in clinical laboratory tests, vital signs, 12lead ECG | throughout the study

SECONDARY OUTCOMES:
Pharmacokinetics and Pharmacodynamics of SB751689 | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site